CLINICAL TRIAL: NCT06328322
Title: Study of Percutaneous Coronary Intervention in Left Main Coronary Artery Disease in Patients With Acute Coronary Syndrome at Sohag University Hospitals
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohammed Bahaa Eldeen Elsayed, assistent lecture- internal medicine -faculty of medicine, Sohag University
Other Study IDs: Soh-Med-24-03-02MD
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Left Main Coronary Artery Disease With Acute Coronary Syndrome
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention in Left Main Artery Disease — To investigate and assess the effectiveness and safety of percutaneous coronary intervention in left main coronary artery disease in sitting of acute coronary syndromes.

SUMMARY:
Acute coronary syndromes (ACS) encompass a spectrum of cardiovascular disorders characterized by the sudden onset of myocardial ischemia. They are primarily caused by atherosclerotic plaque rupture or erosion, leading to partial or complete occlusion of the coronary arteries. Among the various coronary arteries affected, left main coronary artery disease (LMCAD) is of particular concern due to its high anatomical significance and potential for adverse outcomes

The left main coronary artery (LMCA) is responsible for supplying a substantial portion of the left ventricular myocardium, including the interventricular septum and the anterior and lateral walls. Any obstruction or compromise in blood flow within this critical artery can have severe consequences, including myocardial infarction, heart failure, or even sudden cardiac death. The management of LMCAD associated with ACS represents a significant clinical challenge, necessitating prompt and optimal treatment strategies

Among the various coronary arteries affected by atherosclerosis, left main coronary artery disease (LMCAD) holds particular clinical significance due to its anatomical location and the vital role it plays in supplying a substantial portion of the left ventricular myocardium. The left main coronary artery (LMCA) typically bifurcates into the left anterior descending artery (LAD) and the left circumflex artery (LCX), which together provide blood supply to the majority of the left ventricle, including the interventricular septum and the anterior and lateral walls

The selection of an appropriate treatment strategy for LMCAD associated with ACS is a complex decision that requires careful consideration of multiple factors, including patient characteristics, coronary anatomy, severity of ischemia, and procedural expertise. The emergence of several clinical trials and observational studies exploring the efficacy and safety of different revascularization strategies has further complicated the decision-making process

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Acute coronary syndromes (ACS).
* Left main coronary artery disease (LMCAD) on CA.

Exclusion Criteria:

* Patients with contraindications to coronary angiography or invasive procedures.
* Prior history of percutaneous coronary intervention (PCI) with left main stenting.
* Known allergy or intolerance to the medications or devices commonly used during PCI procedures.
* Severe comorbidities or conditions that may limit life expectancy or impact the ability to follow the study protocol.
* Pregnancy or lactation.
* Refusal to participate
* Contra indication to antiplatelet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Age > 18 years.
  * Acute coronary syndromes (ACS).
  * Left main coronary artery disease (LMCAD) on CA.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiac events (MACE) | 6 months post PCI
  cardiovascular death, myocardial infarction, repeat revascularization, and stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Dabrowski EJ, Kozuch M, Dobrzycki S. Left Main Coronary Artery Disease-Current Management and Future Perspectives. J Clin Med. 2022 Sep 28;11(19):5745. doi: 10.3390/jcm11195745. PMID 36233613
- [Background] Waterbury TM, Tarantini G, Vogel B, Mehran R, Gersh BJ, Gulati R. Non-atherosclerotic causes of acute coronary syndromes. Nat Rev Cardiol. 2020 Apr;17(4):229-241. doi: 10.1038/s41569-019-0273-3. Epub 2019 Oct 3. PMID 31582839
- [Background] Spadaccio C, Benedetto U. Coronary artery bypass grafting (CABG) vs. percutaneous coronary intervention (PCI) in the treatment of multivessel coronary disease: quo vadis? -a review of the evidences on coronary artery disease. Ann Cardiothorac Surg. 2018 Jul;7(4):506-515. doi: 10.21037/acs.2018.05.17. PMID 30094215